CLINICAL TRIAL: NCT01404091
Title: Assessment of Nociceptin/Orphanin FQ Peptide Receptor Occupancy After Single Oral Doses of LY2940094 as Measured by Positron Emission Tomography With the Radioligand LY2959530 in Healthy Subjects
Brief Title: A Study of Nociceptin/Orphanin FQ Peptide Receptor Occupancy in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BlackThorn Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14333; I5J-MC-NOAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — LY2940094

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1: 40 milligram (mg) LY2940094 (Experimental): 40 mg LY2940094 was administered orally, one time only (it was originally expected that 100 mg LY2940094 would be administered).
  If the receptor occupancy (RO) for a given dose is lower than 50%, (time to maximum concentration [tmax] or an optimal time window) then a higher dose will be administered to the next cohort whereas if the RO for a given dose is higher than 50%, then a lower dose will be administered to the next cohorts.
  Interventions: Drug: LY2940094
- Cohort 2: 10 mg LY2940094 (Experimental): The dose levels for subjects in Cohort 2 will be defined based on the results of the receptor occupancy (RO) data of previous cohort and the ongoing review of safety data. This dose was determined to be 10 mg, and was administered orally, one time only.
  If the RO for a given dose is lower than 50%, (tmax or an optimal time window) then a higher dose will be administered to the next cohort whereas if the RO for a given dose is higher than 50%, then a lower dose will be administered to the next cohorts.
  Interventions: Drug: LY2940094
- Cohort 3: 4 mg LY2940094 (Experimental): The dose levels for subjects in Cohort 3 will be defined based on the results of the receptor occupancy (RO) data of previous cohort(s) and the ongoing review of safety data. This dose was determined to be 4 mg, and was administered orally, one time only.
  If the RO for a given dose is lower than 50%, (tmax or an optimal time window) then a higher dose will be administered to the next cohort whereas if the RO for a given dose is higher than 50%, then a lower dose will be administered to the next cohorts.
  Interventions: Drug: LY2940094
- Cohort 4: 20 mg LY2940094 (Experimental): The dose levels for subjects in Cohort 4 will be defined based on the results of the receptor occupancy (RO) data of previous cohort(s) and the ongoing review of safety data. This dose was determined to be 20 mg, and was administered orally, one time only.
  If the RO for a given dose is lower than 50%, (tmax or an optimal time window) then a higher dose will be administered to the next cohort whereas if the RO for a given dose is higher than 50%, then a lower dose will be administered to the next cohorts.
  Interventions: Drug: LY2940094

INTERVENTIONS:
Drug: LY2940094 — Administered orally

SUMMARY:
The purpose of this trial is to conduct an assessment of brain nociceptin/orphanin FQ peptide (NOP) receptor occupancy (RO) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index between 19.0 and 30.0 kilogram square meter (kg/m²), inclusive, weight less than 125.0 kilogram (kg), and physical dimensions which appear small enough to fit into the magnetic resonance imaging (MRI) and positron emission tomography scanners (PET)
* Must be in good health, as determined by a medical history, vital signs, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations
* Have venous and arterial access sufficient to allow blood sampling
* Are nonsmokers for at least 3 months prior to Screening, according to self report (meaning zero cigarettes smoked)
* Have a calculated creatinine clearance of greater than (>)70 milliliters per minute (mL/min) at Screening
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

* Male subjects who are not, or whose partners are not willing to use appropriate contraception (condom with spermicidal foam/gel/film/cream/suppository) from the time of the first dose until 3 months after dosing
* Have received any prescribed systemic or topical medication within 14 days of the first dose administration, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety
* Have used any nonprescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration (with the exception of vitamin/mineral supplements) unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety
* Have received any medications, including St. John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety
* Currently enrolled in, have completed, or discontinued within the last 30 days from a clinical trial involving an investigational product or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have donated or lost 50 to 499 mL of whole blood within 30 days, or more than 499 mL whole blood within 56 days preceding first dose administration
* Have a significant history of drug allergy as determined by the Investigator
* Have any clinically significant allergic disease (excluding nonactive hay fever), or any known allergy to LY2940094 as determined by the Investigator
* Have a semi-reclined blood pressure and pulse rate higher than 130/90 millimeters of mercury (mmHg) and 100 beats per minute, respectively, or lower than 90/50 mmHg and 40 beats per minute, respectively
* Consume more than 14 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse/dependence as determined by the Investigator (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 1/6 gill [25 mL] of spirits)
* Have a positive urine drug screen or alcohol breath test result that indicates substance abuse at screening or at admission to any treatment period
* With, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, respiratory, metabolic, endocrine, hematological or other major disorders as determined by the Investigator
* With, or with a history of, any psychiatric illness as assessed with the Symptom Checklist (SCL-90R)
* Have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator
* Have serum hepatitis (B or C), or who are carriers of the hepatitis B surface antigen or hepatitis C antibody, or who have a positive result to the test for human immunodeficiency virus (HIV) antibodies
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risk of participating in the study. In addition, subjects with the following findings will be excluded:

  * Confirmed Bazett's corrected QT interval (QTcB) greater than (>) 450 milliseconds (msec)
  * Bundle branch blocks and other conduction abnormalities (including 2nd or 3rd degree atrioventricular block, complete left bundle branch block, complete right bundle branch block or Wolffe-Parkinson-White syndrome, defined as PR interval less than (<) 110 msec, confirmed by a repeat ECG other than mild first-degree AV block
  * Irregular rhythms other than sinus arrhythmia or occasional rare supraventricular ectopic beats
  * History of unexplained syncope
  * Family history of unexplained syncope or sudden death due to long QT (cardiac output) syndrome
  * T wave configurations are not of adequate quality for assessing corrected QTc intervals
* Have previously completed or been withdrawn from this study or any other study investigating LY2940094
* Subjects who, in the opinion of the Investigator, should not participate in the study
* Taking any excluded medications that cannot be discontinued at admission to the clinical research unit (CRU)
* Have a personal or family history of recurrent seizures or complicated febrile seizures
* Have a history of a significant brain condition/trauma
* Indicates presence of suicidal ideation by answering "yes" to either of the first two questions on the baseline version of the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening
* Have any contraindication to magnetic resonance imaging (MRI) , such as implanted or embedded metal objects or fragments in the head or body that would present a risk during the magnetic resonance imaging (MRI) scanning procedure, or have worked with ferrous metal either as a vocation or hobby (for example, as a sheet metal worker, welder or machinist) in such a way that might have led to unknown, indwelling metal fragments that could cause injury if they moved in response to placement in the magnetic field
* Have had exposure to ionizing radiation in a research study that, in combination with the study tracer, would result in a cumulative exposure that exceeds recommended exposure limits of greater than (>) 20 millisieverts (mSv) in 1 year
* Suffer from claustrophobia and would be unable to tolerate the confined spaces of magnetic resonance imaging (MRI) or positron emission tomography (PET) camera as evidenced by claustrophobia screening
* Without a minimum of 37 inches (112 centimeters [cm] ) from the top of the head to the end of the wrist so as to allow reasonable access to the wrist to take a blood sample during the positron emission tomography (PET) scan
* Have a significant history of hypersensitivity reactions to gelatin capsules.
* Any other condition which, in the opinion of the investigator, would preclude participation in the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Nociceptin/Orphanin FQ Peptide (NOP) Receptor Occupancy at Day 2 | Baseline, Day 2 (occurs 1-4 weeks after baseline)

SECONDARY OUTCOMES:
Pharmacokinetics: maximal plasma concentration (Cmax) of LY2940094 | Predose, up to 29 hours post dose
Pharmacokinetics: area under the concentration- time curve (AUC) of LY2940094 | Predose, up to 29 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario, Canada